CLINICAL TRIAL: NCT00547495
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Tadalafil Administered "On Demand" to Patients With Erectile Dysfunction
Brief Title: Study the Safety and Effectiveness of Tadalafil in Men With Problems Getting or Maintaining an Erection When Taken Prior to Desiring an Erection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5139; H6D-MC-LVDI
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo tablet
  Interventions: Drug: placebo
- 2 (Active Comparator): 5 mg tadalafil
  Interventions: Drug: tadalafil
- 3 (Active Comparator): 10 mg tadalafil
  Interventions: Drug: tadalafil
- 4 (Active Comparator): 20 mg tadalafil
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 5 mg tadalafil tablet, by mouth, as needed, no more than 1 dose per day, for 12 weeks
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: placebo — placebo tablet taken by mouth, as needed, no more than 1 dose per day, for 12 weeks
  Arms: 1
Drug: tadalafil — 10 mg tadalafil tablet, by mouth, as needed, no more than 1 dose per day, for 12 weeks
  Other Names: LY450190; Cialis; IC351
  Arms: 3
Drug: tadalafil — 20 mg tadalafil tablet, by mouth, as needed, no more than 1 dose per day, for 12 weeks
  Other Names: LY450190; Cialis; IC351
  Arms: 4

SUMMARY:
Study to determine how safe and effective tadalafil is for Japanese men taking it when they need to get and keep an erection.

ELIGIBILITY:
Inclusion Criteria:

* 3 months history of erectile dysfunction (ED)
* Anticipate a monogamous relationship with a female sexual partner
* Be able to make minimum required sexual intercourse attempts
* Abstain from using any other ED treatment

Exclusion Criteria:

* Other primary sexual disorders
* History of radical prostatectomy or other pelvic surgery that affected being able to have an erection
* History of penile implant or clinically significant penile deformity.
* Nitrate use
* Certain heart problems

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2004-03; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Effectiveness measured by IIEF score of questions 1-5 and 15 plus the percentages of positive responses to questions 2 and 3 in SEP diary | 12 weeks

SECONDARY OUTCOMES:
Change from baseline to endpoint of various questions from the IIEF and SEP diary | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo, Hokkaido, Japan

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com